CLINICAL TRIAL: NCT00070980
Title: Massage to Enhance Well-Being in HIV-Positive Dominican Children
Brief Title: Massage to Increase Well-Being and Immune Function in Dominican Children Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT001160-01A1 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections; AIDS
Keywords: Complementary Therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Massage

INTERVENTIONS:
Procedure: Massage therapy

SUMMARY:
The purpose of this study is to determine whether massage therapy can improve immune status and enhance well-being in children living in the Dominican Republic who are infected with HIV.

DETAILED DESCRIPTION:
The incidence of pediatric HIV in the Dominican Republic has been rapidly rising, while antiretroviral therapies are not yet readily available to slow disease progression. There is compelling evidence that massage therapy may enhance immune status and alter the course of HIV disease. Increased immune capacity and improvement in HIV disease progression markers have been demonstrated following massage therapy in HIV infected adolescents and adults, even in the absence of antiretroviral treatments. In studies with premature newborns, increased weight gain, decreased stress behavior, and more optimal cognitive and motor development have been reported following massage treatment. This study will examine the efficacy of massage therapy, an affordable and potentially beneficial complementary/alternative treatment, to promote health and enhance well-being in HIV infected children in the Dominican Republic.

Children will be randomly assigned to receive either massage therapy or standard care/friendly visits twice weekly for 12 weeks. Data will be gathered to assess acceptance, safety, and compliance to massage therapy and to examine whether massage treatment has improved immune function, developmental performance, and behavioral function.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Parent/caregiver signature on consent form

Exclusion criteria:

* Unknown HIV status
* Fever, new opportunistic infection, or acute hospitalization within 30 days prior to study entry
* Massage therapy within 30 days prior to study entry
* Unable to have massage (e.g., extensive skin lesions)
* Symptoms of child abuse
* Child born drug-addicted

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54
Dates: Start 2003-03; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Gail Shor-Posner, MD, Principal Investigator — University of Miami
Locations (1):
- CENISMI/Robert Reid Cabral Children's Hospital, Santo Domingo, Dominican Republic